CLINICAL TRIAL: NCT06137547
Title: Hypotension Prediction Index for Prevention of Hypotension During Cardiac Surgery: A Randomized Controlled Trial
Brief Title: HPI for Prevention of Hypotension During Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chun Lin, Attending physician, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20220800015
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery Patients
Keywords: cardiac surgery; hypotension prediction index; hypotension; randomized controlled trial
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI-guided (Experimental): The arterial line of patients in HPI-guided arm will be connected to HemoSphere advanced monitoring platform (EV1000), which will provide HPI value calculated with Acumen Hypotension Prediction Index software.
  Interventions: Device: Hypotension prediction index (HPI)
- non-HPI-guided (No Intervention): The arterial line of patients in non-HPI-guided arm will also be connected to HemoSphere advanced monitoring platform (EV1000) and all hemodynamic parameters will be calculated and showed as HPI-guided arm EXCEPT that the HPI value will not be shown on screen.

INTERVENTIONS:
Device: Hypotension prediction index (HPI) — The hypotension prediction index (HPI) is a value derived from the arterial pressure waveform. It was invented by Edwards Lifesciences through a machine-learning algorithm, and can be calculated with Acumen Hypotension Prediction Index software incorporated in HemoSphere advanced monitoring platform (EV1000). This value, ranging from 0 to 100, predicts the likelihood of a patient trending towards a hypotensive event, which is defined as mean arterial pressure below 65 mmHg for at least one minute.
  Arms: HPI-guided

SUMMARY:
Hypotension prediction index (HPI) was applied in various types of non-cardiac surgery with convincing benefits of preventing hypotensive events and clinical sequelae. Although HPI was validated in cardiac surgery, its clinical benefits are not proven yet. We aim to evaluate its effects on intraoperative hypotension and postoperative adverse events in cardiac surgery. In this randomized, single-blind trial, we will enroll adults scheduled for elective primary cardiac surgery under general anesthesia. Participants will be randomly assigned to intraoperative HPI-guided or non-HPI-guided hemodynamic management. The primary endpoint is the time-weighted average intraoperative hypotension below a mean arterial pressure threshold of 65 mmHg. The secondary endpoints are postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* adult
* elective, primary, isolated coronary arterial bypass surgery (CABG) or isolated valve surgery
* provide inform consent.

Exclusion Criteria:

* arrhythmia (e.g., atrial fibrillation, atrial flutter)
* intracardiac shunts
* preoperative inotropic usage
* preoperative supportive devices usage (e.g., intra-aortic balloon pump, extracorporeal membrane oxygenation, left ventricular assist device, or right ventricular assist device)
* receiving urgent or emergent procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
TWA (time-weighted average) of intraoperative hypotension | From induction to the end of surgery. (If cardiopulmonary bypass (CPB) is adopted, the time of CPB will not be counted in)
  Time-weighted average of intraoperative hypotension below 65 mmHg

SECONDARY OUTCOMES:
incidence of hypotension | from induction to the end of surgery (excluding CPB time)
duration of hypotension | from induction to the end of surgery (excluding CPB time)
postoperative complications | after surgery until discharge, assessed up to 30 days
  including acute kidney injury, arrhythmia, myocardial infarction determined by levels of cardiac enzymes, stroke, and mortality
length of ICU stay | after surgery until ICU discharge, assessed up to 30 days
length of hospital stay | after surgery until hospital discahrge, assessed up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay memorial hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not understand the individual patient data (IPD) sharing platform through enough.